CLINICAL TRIAL: NCT02135094
Title: Short Term Effects of Long Duration Low Intensity Continuous Ultrasound for Trapezius Muscle Pain
Brief Title: Low Intensity Ultrasound Therapy for Upper Back Pain Relief
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZetrOZ, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TP-02; 201306603 (Other: Schulman Associates IRB)
Record Dates: First submitted 2014-05-02; First posted 2014-05-09 (Estimated); Results first posted 2018-06-11 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Muscle Spasm
Keywords: trapezius; upper back; muscle pain; pain relief; ultrasound; double blind; Sam; ZetrOZ; muscle; LITUS; low intensity therapeutic ultrasound
MeSH Terms: conditions — Spasm; Myalgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active ultrasound therapy device (Experimental): Patients receive treatment from the Sam Ultrasonic Diathermy Device for 4 hours on days when their trapezius muscle pain score is at least a 3 on a scale of 0-10 (NRS). The active device emits continuous ultrasound at 3 megahertz (MHz) frequency and 0.132 watts/cm2 intensity
  Interventions: Device: Active ultrasound therapy device
- Placebo ultrasound therapy device (Placebo Comparator): Patients apply the Sam Ultrasonic Diathermy Device for 4 hours on days when their trapezius muscle pain score is at least a 3 on a scale of 0-10 (NRS). The placebo device appears and operates identically to the active device except that it does not emit ultrasound.
  Interventions: Device: Placebo ultrasound therapy device

INTERVENTIONS:
Device: Active ultrasound therapy device — low intensity continuous therapeutic ultrasound at 3 megahertz (MHz) frequency and 0.132 Watts/cm2 for treatment duration of 4 hours per day
  Other Names: ZetrOZ ultrasound device; wearable ultrasound device; long duration ultrasound; LITUS device; long duration low intensity device
  Arms: Active ultrasound therapy device
Device: Placebo ultrasound therapy device — The placebo device appears and operates identically to the active device except that it does not emit ultrasound.
  Other Names: ZetrOZ ultrasound device; wearable ultrasound device; long duration ultrasound; LITUS device; long duration low intensity device
  Arms: Placebo ultrasound therapy device

SUMMARY:
The purpose of this study is to measure the effectiveness of a wearable therapeutic ultrasound device for relief of pain associated with the trapezius muscle of the upper back over a 4-week period. The trapezius muscle is a wide, flat, superficial muscle that covers most of the upper back and the posterior of the neck.The hypothesis is that the ultrasound device will lower the reported daily pain level of subjects suffering from trapezius muscle pain in their upper back.

Subjects who participate in the study will self-administer the ultrasound device daily if pain is rated 3.0 or higher on the numeric rating scale (0-10). Subjects will be required to visit the clinical site at enrollment and weeks 2 and 4 for a total of 3 visits. Subjects will report their daily pain levels in a diary. Subject will also report pain levels at 30 min, 2 hours, and 4 hours (treatment completion) after start of each treatment.

The wearable ultrasound device, Sam®, has been cleared by the FDA for pain relief, relief of joint contracture, relief of muscle spasm, and increased circulation.

DETAILED DESCRIPTION:
The study will have approximately 33 subjects randomly assigned into a user group (active ultrasound device) of 25 participants or a control group (inactive ultrasound device) of 8 participants with an equal number of males and females in each group. The research coordinator will be blinded to the assignment of devices to each group.

The daily pain scores reported by patients who receive active devices will be compared to those who receive placebo devices.

Background:

Approximately 50 to 80 million people in the United States suffer from some form of chronic pain. Back pain is the most common neurological disorder in the United States after headaches and costs consumers nearly $50 billion annually. Pharmaceuticals currently dominate the treatment options despite a myriad of public health problems including cost, untoward side effects, and addiction to widely available opioid analgesics. Non-pharmaceutical treatments, such as the one under test, provide a safer and potentially lower cost alternative to traditional analgesic use.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 65 years.
* Has acute trapezius muscle pain that has been assessed by a health care practitioner.
* Has a NRS pain severity score of 3.0 or higher in the trapezius muscle 3-4 times over the past week prior to enrolling in the trial.
* Subjects must be willing and able to self-administer treatment daily within their place of residence or during normal daily activity, excluding bathing, showering, or other water activities which may result in submersion of the device under test.
* Not taken any prescription pain medications or muscle relaxers in the 5 days prior to the study and agree not to take any during the study and to maintain any dosage of NSAIDs (nonsteroidal antiinflammatory drug) or non-prescription pain medications constant during the study
* Has access to a mobile phone or camera and the help of another individual to take a picture of the upper back area immediately after use of the device

Exclusion Criteria:

* Subjects with known neuropathy will be excluded from the study
* Women who are pregnant may not participate.
* Prisoners
* Smokers
* Subjects with Type I or Type II Diabetes
* Subjects who have had surgery in the target area within the last 6 months will be excluded from the study.
* Subjects who are non-ambulatory (i.e. who cannot walk) will be excluded from the study.
* Subjects who refuse to agree to not increase current use or initiate new use of pain medication during the course of the trial unless medically necessary to ensure patient safety.
* Subjects who refuse to agree to not use any cream, gel, or topical solution during the administration of treatment other than the approved ultrasound gel provided to the subject at the initiation of the study.
* Subjects who refuse to discontinue massage therapy or spinal manipulation during the duration of this study.
* Subjects who have had massage therapy within 1 day of beginning the protocol
* Subjects who refuse to discontinue all other interventional treatment modalities (i.e. transcutaneous electrical nerve stimulation (TENS), ultrasound)
* Subjects who had a local corticosteroid or PRP (platelet-rich plasma) injection within the past 3 months.
* Subjects who have a clinically significant or unstable medical or psychological conditions that would compromise participation in the study.
* Subjects who have participated in another clinical trial for an investigational drug and/or agent within 30 days prior to screening.
* Subjects involved in any injury-related litigation in the target area.
* Subjects with abnormal neurological history, lumbar radicular symptoms, spinal stenosis, foot drop, herniated nucleus pulposus (gel-like substance within a spinal disc), or other structural defects.
* Subjects with back pain related to major trauma in the last 6 months
* Subjects with open sores or wounds in the treatment area that would prevent use of the device

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George K. Lewis, PhD, Principal Investigator — ZetrOZ, Inc.
Locations (1):
- ZetrOZ, Inc., Trumbull, Connecticut, United States

REFERENCES:
- [Derived] Petterson S, Plancher K, Klyve D, Draper D, Ortiz R. Low-Intensity Continuous Ultrasound for the Symptomatic Treatment of Upper Shoulder and Neck Pain: A Randomized, Double-Blind Placebo-Controlled Clinical Trial. J Pain Res. 2020 Jun 2;13:1277-1287. doi: 10.2147/JPR.S247463. eCollection 2020. PMID 32606899

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Ultrasound Therapy Device | Placebo Ultrasound Therapy Device
Started | 25 | 8
Week 2 | 25 | 8
Week 3 | 25 | 8
Week 4 | 25 | 8
Completed | 25 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Ultrasound Therapy Device | Placebo Ultrasound Therapy Device | Total
Number analyzed (Participants) | 25 | 8 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.2 (13.9) | 30.3 (10.9) | 33.3 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 5 | 21
  Male | 9 | 3 | 12
Region of Enrollment [Number; unit: participants]
  United States | 25 | 8 | 33
Height [Mean (Standard Deviation); unit: cm] | 169.8 (12.1) | 169.1 (9.7) | 169.6 (11.4)
Weight [Mean (Standard Deviation); unit: kg] | 75.1 (13.1) | 72.2 (22.4) | 74.4 (15.0)

OUTCOME MEASURES:

1. Primary Outcome: Pain on the Numeric Rating Scale (NRS)
Description: Patients applied the ultrasound device when trapezius muscle pain exceeds a score of 3 or higher by numeric rating scale (NRS). NRS range was 0-10 with 0 being no pain and 10 the worst pain possible. Device maybe be worn safely for 4 h per day for 7 days a week. Participants recorded NRS score daily (pre-treatment) and on days when the device was applied participants recorded pain 30 minutes into treatment, 2 hours into treatment and post-treatment (after 4 hours). The post-treatment score is used to find the week average and standard deviation.
Time Frame: Week 1, Week 2, Week 3, Week 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Ultrasound Therapy Device | Placebo Ultrasound Therapy Device
Number analyzed (Participants) | 25 | 8
units on a scale
  Week 1 | 5.60 (1.58) | 5.44 (1.95)
  Week 2 | 3.54 (1.64) | 4.58 (2.20)
  Week 3 | 3.09 (1.54) | 3.92 (2.10)
  Week 4 | 2.98 (1.62) | 3.86 (2.30)

2. Primary Outcome: Pain on the Numeric Rating Scale (NRS) Change From Day 1 Pre-treatment.
Description: The Day 1 pre-treatment score was used to find the change in pain each week, rated on the numeric rating scale (NRS). NRS was rated from 0-10 with 0 being in no pain and 10 the worst pain possible. Weekly averaged post-treatment scores were subtracted from Day 1 pre-treatment score.
Time Frame: Day 1 through Week 1, Week 2, Week 3, and Week 4
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active Ultrasound Therapy Device | Placebo Ultrasound Therapy Device
Number analyzed (Participants) | 25 | 8
units on a scale
  Week 1 Change from Day 1 | -2.05 [-2.76 to -1.35] | -0.860 [-2.53 to 0.810]
  Week 2 Change from Day 1 | -2.34 [-3.03 to -1.65] | -0.693 [-2.49 to 1.11]
  Week 3 Change from Day 1 | -2.51 [-3.18 to -1.83] | -1.52 [-3.14 to 0.110]
  Week 4 Change from Day 1 | -2.61 [-3.34 to -1.90] | -1.58 [-3.40 to 0.24]

3. Secondary Outcome: Pain on the Numeric Rating Scale Assessed Before, During, and After Treatment.
Description: Participants recorded pain rated on the numeric rating scale (NRS) at 4 time points: before treatment, 30 minutes into treatment, 2 hours into treatment, and directly after treatment. NRS range was from 0-10 with 0 being no pain and 10 the worst pain possible. The average time point scores across the study is used to assess pain during treatment.
Time Frame: Day 1 through Week 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Ultrasound Therapy Device | Placebo Ultrasound Therapy Device
Number analyzed (Participants) | 25 | 8
units on a scale
  Before Treatment | 5.40 (1.50) | 5.22 (2.14)
  30 minutes into Treatment | 4.99 (1.39) | 4.98 (2.13)
  2 hours into Treatment | 4.04 (1.45) | 4.61 (2.08)
  Post-treatment | 3.24 (1.61) | 4.34 (2.26)

4. Secondary Outcome: Change in Pain Rated on Numeric Rating Scale (NRS) From Pre-treatment to 30 Minutes Into Treatment, 2 Hours Into Treatment, and Post-treatment (4 Hours Into Treatment)
Description: The numeric rating scale (NRS) was used to assess pain before treatment, 30 minutes into treatment, 2 hours into treatment, and post-treatment. NRS range was from 0-10 with 0 being in no pain and 10 the worst pain possible. Change in pain was calculated by subtracting intra-treatment and post-treatment average scores from pre-treatment average score.
Time Frame: Day 1 through Week 4
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active Ultrasound Therapy Device | Placebo Ultrasound Therapy Device
Number analyzed (Participants) | 25 | 8
units on a scale
  Pain score change after 30 minutes | -0.416 [-0.599 to -0.218] | -0.237 [-0.713 to 0.239]
  Pain score change after 2 hours | -1.36 [-1.55 to -1.16] | -0.615 [-1.09 to -0.145]
  Pain score change after 4 hours | -2.16 [-2.36 to -1.95] | -0.885 [-1.37 to -0.394]

5. Secondary Outcome: Comparison of Pain Level Using Global Rating of Change (GROC) Scale.
Description: Participants were asked to report how their body feels overall compared to the day before, on days when the ultrasound device (or placebo) were applied. The score was reported after the 4-hour treatment completion and rated on a 15-point global rating of change scale, with -7 being "a very great deal worse" than the day before, 0 being "no change" from the day before, and +7 being "a very great deal better" than the day before. The weekly average GROC and average GROC for the entire study (Overall) were assessed.
Time Frame: Week 1, Week 2, Week 3, Week 4, Overall
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Ultrasound Therapy Device | Placebo Ultrasound Therapy Device
Number analyzed (Participants) | 25 | 8
units on a scale
  Week 1 | 2.35 (1.96) | 0.76 (1.89)
  Week 2 | 2.84 (2.01) | 0.53 (2.44)
  Week 3 | 3.21 (2.45) | 0.36 (1.99)
  Week 4 | 3.09 (2.37) | 0.14 (1.93)
  Overall | 2.84 (2.21) | 0.46 (2.08)

ADVERSE EVENTS:
Arm/Group | Active Ultrasound Therapy Device | Placebo Ultrasound Therapy Device
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/8
Other Adverse Events (participants affected / at risk) | 0/25 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No